CLINICAL TRIAL: NCT03511716
Title: HRT Observational Study of a Mitral Bridge in Patients With Moderate to Severe Mitral Valve Regurgitation to Evaluate Device Safety and Performance
Brief Title: Observational Study of the Heart Repair Technologies Mitral Bridge in Treating Mitral Valve Regurgitation
Acronym: HRT
Status: Terminated | Type: Observational
Why Stopped: Could not enroll enough patients and ran out of $$ to manufacture more devices
Sponsor: Heart Repair Technologies, Inc. (Industry)
Collaborators: Na Homolce Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HRT Mitral Bridge
Record Dates: First submitted 2018-04-09; First posted 2018-04-30 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2019-08

CONDITIONS: Mitral Regurgitation
Keywords: Mitral Insufficiency; Mitral Valve Incompetence
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: HRT Mitral Bridge Mitral Valve Repair — Surgical mitral valve implant intended to reduce mitral regurgitation by direct reduction of the septo-lateral mitral annular diameter, promoting early coaptation of the valve leaflets and restraining the leaflets below the intra-annular plane

SUMMARY:
Prospective, observational, multi-center trial in which patients with mitral regurgitation sufficient to merit mitral valve repair will receive a surgical transvalvular, intra-annular Mitral Bridge™ to reduce or eliminate mitral regurgitation.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and performance of the Mitral Bridge device in the correction of mitral valve regurgitation in patients who qualify for mitral valve repair as defined by the American Society of Echocardiography (ASE). The device is a single use, mitral valve implant designed to reduce mitral regurgitation by reducing the septo-lateral mitral annular diameter, promoting early coaptation of the valve leaflets and restraining the leaflets below the intra-annular plane.

The protocol was designed as a First In Man (FIM) with a 6-month follow up but was amended to follow the enrolled patients for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients moderate to severe, symptomatic functional (ischemic or dilated cardiomyopathies) mitral regurgitation or mitral regurgitation caused by dilation of the mitral annulus who qualify for mitral valve repair with cardiopulmonary bypass
* Mitral regurgitation must meet the following criteria:
* The primary regurgitant jet is central, originating from mal coaptation of anterior and posterior leaflets of the mitral valve.
* If a secondary jet is present, the jet must be considered clinically insignificant.
* Women of child-bearing potential have a negative pregnancy test

Exclusion Criteria:

* Evidence of severe mitral annular and leaflet calcification.
* Patient is hemodynamically unstable.
* Patient has hypertrophic cardiomyopathy and has systolic anterior motion of the leaflets.
* Patient requires emergency surgery.
* Patient has echocardiographic evidence of endocarditis or rheumatic heart disease.
* Transesophageal Echocardiogram (TEE) is contraindicated or cannot be performed intraoperatively for any reason.
* Patient has known chronic, dialysis-dependent renal failure.
* History of stroke, transient ischemic attack (TIA) or reversible ischemic neurological disease within the last three (3) months.
* History of gastrointestinal bleeding within the last three (3) months.
* History of hypersensitivity or allergy to aspirin
* History or hypersensitivity to clopidogrel (Plavix) or its congeners.
* Active or treated malignancies in the last twelve (12) months.
* Patient is participating in another clinical study for which follow-up is currently ongoing.
* Women of child-bearing age who have not had a negative pregnancy test.
* Patient with non-cardiac co-morbidities and life expectancy < 1 year.
* Patient has a condition that, in the opinion of the Investigator, precludes participation, including willingness to comply with all follow-up procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 21 with moderate to severe, functional (ischemic or dilated cardiomyopathies) mitral regurgitation or mitral regurgitation caused by dilation of the mitral annulus who qualify for mitral valve repair
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical Success | One, 3, 6,12, 24, 36, 48, and 60 months
  - Freedom from subsequent open mitral valve repair or replacement

SECONDARY OUTCOMES:
Preservation or improvement of left ventricular remodeling | One, 3, 6,12, 24, 36, 48, and 60 months
  Change in Left Ventricular status
Preservation of improvement in NYHA (New York Heart Association) functional class. | One, 3, 6,12, 24, 36, 48, and 60 months
  Change in NYHA (New York Heart Association) functional class.

CONTACTS AND LOCATIONS:
Overall Officials: Štěpán ČERNÝ, MD, PhD, MBA, Principal Investigator — Cardiac Surgeon, Head of Hybrid Operating Room,
Locations (1):
- Na Homolce Hospital, Prague, Homolka, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cerny S, Benesova M, Skalsky I, Patel NC, Subramanian VA. Persistent reduction of mitral regurgitation by implantation of a transannular mitral bridge: durability and effectiveness of the repair at 2 years-results of a prospective trialdagger. Eur J Cardiothorac Surg. 2019 May 1;55(5):867-873. doi: 10.1093/ejcts/ezy423. PMID 30590416